CLINICAL TRIAL: NCT06732453
Title: Adaptation of the Yoga Skills Training for Relief of Nausea and Vomiting in Patients With Functional Dyspepsia and Gastroparesis
Brief Title: Brain-Gut Yoga for Functional Dyspepsia and Gastroparesis (FD-GP)
Acronym: FD-GP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00122246; 400983697 (Other: American Neurogastroenterology and Motility Society)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: Functional Dyspepsia; Gastroparesis
Keywords: Yoga; Disorders of the upper gastrointestinal (GI) tract; Brain-gut behavior
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seated Yoga Intervention (Experimental): Two one-hour yoga sessions with home practice administered individually by a yoga interventionist in GI clinic
  Interventions: Other: Seated Yoga Skills Training in Functional Dyspepsia and Gastroparesis (FD-GP)

INTERVENTIONS:
Other: Seated Yoga Skills Training in Functional Dyspepsia and Gastroparesis (FD-GP) — Two one-hour chair-based yoga sessions that will include gentle movements, breathing practices, and meditation, along with home practice.

SUMMARY:
The purpose of this research study is to assess whether using a yoga-based intervention in practice is feasible (possible) and acceptable to patients with Functional Dyspepsia and/or Gastroparesis (FD-GP).

DETAILED DESCRIPTION:
This research looks to adapt an existing seated yoga intervention, designed for patients with GI cancer, for testing in patients with disorders of the upper GI tract by conducting a field test with FD-GP patients to assess feasibility and acceptability and refine the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Functional Dyspepsia or Gastroparesis (FP or GP) diagnosed by a physician using standard criteria
* Signed, written consent

Exclusion Criteria:

* Co-morbid Gastrointestinal or related disorders documents in the medical record: celiac disease, inflammatory Bowel Disease(active), gastrointestinal obstruction (if current in the last 6 months), any GI surgery within the last 6 months), chronic pancreatitis or any pancreatic or biliary disease, cirrhosis or any chronic liver disease other than metabolic associated hepatic disease (MASH), any malignancy (except skin cancer already resected and surgically in remission)
* A positive screen for the following: current psychotic symptoms, elevated suicide risk, active eating disorder, cognitive impairment, current harmful alcohol or substance use
* Does not understand English
* Underwent a regular yoga or other mediative movement practice (tai chi or qi gong) in the past 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Screening Rate | Week 0
  Tracking the number of screened participants, those who are eligible, and the percent who agree to participate.
Recruitment Rate | Week 0
  Total number of patients who enrolled and proportion of patients eligible who enrolled
Retention Rate | Week 2
  Total number of participants who enrolled in the study who remained until completion
Adherence Rate | Week 2
  Completion of 75% of the planned in-person sessions will be considered adherent; home practice will be tracked via daily logs sent back to study team electronically.
Assessment Process Time | Week 2
  Amount of time needed for assessments.
Acceptability of Intervention Score | Week 2
  Overall acceptability of intervention. Target acceptability ratings of at least 4 (agree/completely agree) on a scale of 1 to 5, with a score of 5 being the most acceptable.
Client Satisfaction Questionnaire Score | Week 2
  Assesses satisfaction with treatment. Scores range from 8 to 32; higher scores indicate more satisfaction.
Intervention Usability Scale Score | Week 2
  Measures intervention usability. Scores range from 0-100; a score of 70 or greater may be considered adequate.
Visual analog scale for pain (VAS) score | Week 1, Week 2
  Acute effects using a VAS scale of nausea and psychological distress ranging 0 (none at all) to 100 (as much as there could be) before and after each session to assess immediate relief of symptoms. Higher scores indicate more nausea and psychological distress.
Semi-Structured Interview | Week 2
  30-minute qualitative interview for perspectives on the barriers and facilitators to program engagement and suggestions for improvement, benefits of yoga intervention, and specific questions about format, usability, and burden of the intervention and current and future assessments. Key domains corresponding to the research goals will be developed based on the interview guide. All responses within each domain will be summarized to identify key findings which will be used to inform adaptation of the intervention.
Semi-Structured Interview | Week 3
  30-minute qualitative interview for perspectives on the barriers and facilitators to program engagement and suggestions for improvement, benefits of yoga intervention, and specific questions about format, usability, and burden of the intervention and current and future assessments. Key domains corresponding to the research goals will be developed based on the interview guide. All responses within each domain will be summarized to identify key findings which will be used to inform adaptation of the intervention.
Semi-Structured Interview | Week 4
  30-minute qualitative interview for perspectives on the barriers and facilitators to program engagement and suggestions for improvement, benefits of yoga intervention, and specific questions about format, usability, and burden of the intervention and current and future assessments. Key domains corresponding to the research goals will be developed based on the interview guide. All responses within each domain will be summarized to identify key findings which will be used to inform adaptation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Thakur, MD, Principal Investigator — Wake Forest University
Locations (1):
- Atrium Health Gastroenterology and Hepatology Kenilworth, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No